CLINICAL TRIAL: NCT04764916
Title: Prospective Evaluation of Exparel Adductor Canal Field Block for Pain Control After Anterior Cruciate Ligament Reconstruction
Brief Title: Evaluation of Exparel Adductor Canal Field Block for Pain Control After ACL Reconstruction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-574
Record Dates: First submitted 2021-02-01; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Anterior Cruciate Ligament Tear; Pain, Postoperative; Opioid Use
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: One study group receives standard bupivacaine. One group receives liposomal bupivacaine (Exparel). All other study procedures are identical
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Surgeons and patients will be blinded to study arm until 2 week post-operative visit. Anesthesiology and their staff will not be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exparel/Intervention group (Experimental): Will receive 10mL of standard 0.5% bupivacaine followed by 10mL of liposomal bupivacaine as adductor canal field block preoperatively
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacaine Hydrochloride
- Standard of Care group (Active Comparator): Will receive 20mL of standard 0.5% bupivacaine as adductor canal field block preoperatively
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Liposomal bupivacaine — Liposomal bupivacaine will be used as adductor canal block
  Arms: Exparel/Intervention group
Drug: Bupivacaine Hydrochloride — This is the facility's standard of care medication for this procedure

SUMMARY:
This is a prospective, randomized study for adult patients presenting to the Carilion Clinic Institute of Orthopedics and Neurosurgery. Patients undergoing isolated ACL reconstruction will be eligible for inclusion. All patients will receive an adductor canal block (either with bupivacaine or Exparel. Patients will be given a pain diary for self-report of pill counts, pain scores, block duration, and pain control satisfaction). Pill counts and pain scores will also be taken by a team member at two and six-week post-operative visits. Primary outcomes include opioid requirements and pain scores.

DETAILED DESCRIPTION:
Patients who have an isolated anterior cruciate ligament reconstruction scheduled to be performed at Roanoke Ambulatory Surgery Center (RASC) by one of the participating Carilion surgeons will be prescreened, assessed for eligibility and consented at the pre-operative visit.

This office visit already includes: a formatted discussion regarding the risks, benefits and alternatives to surgery; and a review of the opioid policy and patient agreement used by Carilion Clinic's Institute for Orthopaedics and Neurosciences (ION). The PI or sub-investigators will conduct the discussion regarding the rationale and use of adductor canal block (ACB) with the procedure, the rationale for assessment of alternate medications used for the study, and any other pertinent details. An approved research team member will review all sections of the IRB approved research consent in detail, in person at the pre- operative visit. All questions will be answered, and physical signatures will be obtained. Both research groups, control and experimental, will sign the same consent document. A copy of the signed consent will be provided to the participant.

All participants will be given a pain diary to take home and begin filling out on post-op day #1 (POD#1). Per patient preference, pain diary may be physical copy or done electronically via REDCap.

All participants will be instructed on how to record entries in the pain diary by an approved research team member, and will be instructed to record entries daily. The pain diary will have templated pages with areas to record the amounts and names of medications they consumed, Numeric Rating Scale (NRS) score, Intervention Based Pain Scale (IBPS) score, as well as satisfaction levels and a place to record how long their anesthetic block lasted. NRS responses will be indicated by circling a number ranging from 0 (no pain) to 10 (worst pain imaginable). IBPS responses will be indicated by asking patients to check a box next to the statement that best describes their pain management that day. A numerical score will be associated with responses ranging from 1-6. Patient satisfaction will be asked regarding their pain management for the day on a 5-point likert scale ranging from very dissatisfied to very satisfied. Field block duration will be recorded in hours.

All participants will be provided the same information and education regarding postoperative pain management protocol and expectations.

This is standard of care at Carilion Clinic's ION and includes:

A review of the opioid policy and patient agreement used by Carilion Clinic's ION as well as a discussion about proper use of the pain medication to be prescribed for postoperative pain management A discussion regarding the pain blocks used with the procedure and their likely duration of analgesia A discussion of scheduled postoperative visits and how to contact the office with questions/concerns regarding recovery

The random number generator feature in REDcap will be used to randomly assign subjects to receive the standard Bupivacaine HCl ACB or the Exparel ACB. Surgery schedules at RASC are released on Friday the week before. We will retrieve the surgery schedule on Fridays from RASC, find our study subjects, and randomize them to group A (Exparel) or group B (Bupivacaine HCl) that same day (the Friday before surgery). Once the subjects are randomized, we will communicate the randomization to a RASC staff member, and they will put the arm designation (group A or group B) in an envelope and attach it to the subject's chart for the day of surgery. The contents of the envelope will only be seen by Anesthesia providers and charge nurses prior to the surgery with no other study staff in the room (so the blind is not broken). Charge nurses and anesthesiologists at RASC will be unblinded to the definitions of groups A & B in order to gather and administer the proper medications. Charge nurses will see the designation of group A or B in the envelope attached to the subject's chart and gather the appropriate anesthetic medications for the anesthesiologists. Surgeons will not be in the room at the time of anesthetic administration. The patient and all other providers including physicians and physician assistants will be blinded to the result of the randomization. Patients may opt to be unblinded to their group assignment at their 6- week post- operative visit.

All patients will be undergoing a routine ACLR. The procedure will not deviate from the standard of care operation that is typically performed. All patients will receive post-operative pain medication regimens established by the participating physicians. This regimen is as follows: Loading dose of Toradol in OR (15- 30mg dependent on patient risk factors) followed by prescription for 20 tabs oral Hydrocodone /Acetaminophen (Norco) 5/325 mg and 15 tabs oral Toradol 10mg. Intraoperative supplemental anesthesia will include Marcaine 0.5% or 1% with epinephrine (dependent on medication availability). Additional NSAID use and DVT prophylaxis will be left to discretion of patient and provider.

Prior to their operation, all patients will receive an ultrasound-guided ACB by a pool of anesthesia providers at RASC. The only difference between subject groups is that the control group will receive a standard Bupivacaine HCl ACB and the experimental group will receive an Exparel ACB.

On the day of surgery all patients will be brought to the pre-operative holding area at RASC where they are seen prior to the surgical procedure by both the operating surgeon and the anesthesiologist. The operating surgeon will review the surgical procedure with all patients and will mark the side and location of the procedure. The anesthesiologist will review the ACB procedure with the patient and ensure correct side and location marked by physician. Before the anesthesiologist begins administration of the ACB, a surgical time-out is performed with the operating surgeon, the anesthesiologist and the patient. This is a universal procedure and is the final reassurance of accurate patient identity, surgical site, and planned procedure. In addition, the correct patient positioning, presence of allergies, and the availability of relevant documents and diagnostic tests, instruments, implants and other pertinent equipment are confirmed during this time. A second time-out will also be performed prior to the start of the operation.

In the pre-operative holding area, the anesthesiologist will administer the ACB under ultrasound guidance. Patients in the control group will receive 20mL of standard 0.5% bupivacaine. Patients in the intervention group will receive 10mL of standard 0.5% bupivacaine, followed by 10mL of Exparel. If patients are unable to sit still during ACB administration, they may be sedated by the anesthesiologist with one of the following (Medications and dosages vary based on patient need. Most common medications used listed below):

Versed Fentanyl Propofol

15-20 minutes after administration of ACB's (Bupivacaine HCl or Exparel), all patients will undergo induction of anesthesia by the anesthesiologist. After general anesthesia takes effect, all patients will be operated on by their orthopaedic surgeon.

All participants will be called or seen in the office within 72 hours after surgery to assess pain status, ensure adequate pain management, and will be reminded to complete the pain diary.

All participants will fill out a pain diary during the first 2 weeks post-operatively that will assess 5 measures:

Medication consumption (dose & number of pills) - will be asked to record daily Pain score on the NRS - will be asked to record daily Pain score on an institutional IBPS - will be asked to record daily Patient satisfaction - will be asked to record daily Block duration - will be reminded to record if their block has worn off, and if so, how many hours it was effective (until they regained sensation).

All participants will be called before their 2- and 6-week follow-up appointments and will be asked to bring in their pain diaries as well as their opioid medication pill bottles to their visit so that pill counts may be conducted.

All calls will be made by trained, authorized site delegates. There will be a locked drop-box in the ION building where patients can drop off their pain diaries after their 2-week follow- up appointment if they forget to bring it in to their appointment.

All participants will come into the office for a follow-up appointment at 2-weeks and all particpants will have either a telehealth or in-person appointment at 6 weeks. 2-week appointments will be in-person, as they will need to come in for suture removal.

At the first follow up appointment (week 2), all participants will be expected to bring in their opioid medication pill bottles and their pain diaries per instructions given at study enrollment and on the reminder phone call. All participants will be shown where the lock boxes are to deposit their pain diaries. Pill counts will be conducted and recorded as well as number of refills.

At the second follow up appointment (week 6), all participants will be expected to bring in their opioid medication pill bottles (if in person) per instructions given at study enrollment and on the reminder phone call.

Pill counts will be conducted and recorded as well as number of refills. If 6-week visit is done via telehealth, the same procedures will apply accordingly.

All participant follow-up appointments will be conducted at Carilion's Institute for Orthopaedics and Neurosciences (ION) or via telemedicine, and should not take significantly longer than normal follow up appointments. Slightly increased visit duration related to conducting pill counts should not exceed about 5 minutes. All participants will be enrolled in the study for 6 weeks after their surgical date, at which point their involvement in the study will conclude.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Presenting to Carilion Clinic Institute of Orthopedics and Neuroscience
* Receiving an isolated, first-time ACL reconstruction
* Operation to be performed at the Roanoke Ambulatory Surgery Center

Exclusion Criteria:

* Prior opioid use within 30 days of operation
* Under 18 or over 65 years old
* Use of opioids for chronic pain management
* Patients with multi-ligament injuries
* Patients who are receiving a revision of a previously reconstructed ACL
* Patients with an allergy to the study drug(s)
* Patients not medically eligible for surgery
* Women who are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-02-16 (Estimated); Study Completion 2022-03-02 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | 2 weeks post-operatively
  Total amount of opioids taken by each patient
Total opioid consumption | 6 weeks post-operatively
  Total amount of opioids taken by each patient

SECONDARY OUTCOMES:
Pain control quantified by numerical rating scale | 2 weeks post-operatively
  Pain control reported by patient uses NRS pain scale. 0-10 with 10 being worst pain.
Pain control quantified by intervention-based pain scale | 2 weeks post-operatively
  Pain control reported by patient using our intervention-based pain scale. 1-6 with 6 being most difficult to control pain.
Block length | Self reported anytime from immediately post-op until 2 weeks post-operatively. Likely 1-3 days
  Duration of adductor canal block, reported by patient

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Miller, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic Institute for Orthopaedics and Neurosciences, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No